CLINICAL TRIAL: NCT03598218
Title: A Multicenter, Prospective, Randomized, Phase II Trial Evaluating Hypofractionated Versus Conventionally Fractionated Radiotherapy for Initial Distant Metastases Nasopharyngeal Carcinoma
Brief Title: Hypofractionated Versus Conventionally Fractionated Radiotherapy for Initial Distant Metastases Nasopharyngeal Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wei Jiang (Other)
Collaborators: Wuzhou Red Cross Hospital (Other); Guangxi Naxishan Hospital (Other); Nanning Monority Hospital (Unknown); Lingshan people's Hospital (Unknown)
Responsible Party: Sponsor-Investigator, Wei Jiang, Wei Jiang, MD, PhD, Guilin Medical University, China
Organization: Guilin Medical University, China (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GLMU-03
Record Dates: First submitted 2018-07-14; First posted 2018-07-26 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Hypofractionated Radiation; initial distant metastases; nasopharyngeal carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypofractionated dose IMRT (Experimental): Patients receive hypofractionated with a low total dose radiation with induced chemotherapy and adjuvant chemotherapy.
  Interventions: Radiation: Hypofraction radiation
- Standard-dose IMRT (Experimental): Patients receive standard-dose radiation therapy with induced chemotherapy and adjuvant chemotherapy..
  Interventions: Radiation: Standard dose IMRT

INTERVENTIONS:
Radiation: Hypofraction radiation — Hypofractionated dose IMRT: GTVnx 60Gy, GTVnd 60Gy, PTV1 50Gy and PTV2 45Gy in 25 fractions, 5 days/week.
  Induced chemotherapy: Paclitaxel 135mg/m2 D1+Cisplatin 80mg/m2 D1(or D1-3), 3-week chemotherapy for 3 cycles. After radiation, patients receive adjuvant chemotherapy Paclitaxel 135mg/m2 D1+Cisplatin 80mg/m2 D1(or D1-3), 3-week chemotherapy for 3 cycles.
  Arms: Hypofractionated dose IMRT
Radiation: Standard dose IMRT — Standard dose IMRT: GTVnx 69.69Gy, GTVnd 60-68Gy, PTV1 54.9Gy and PTV2 54Gy in 33 fractions, 5 days/week.
  Induced chemotherapy: Paclitaxel 135mg/m2 D1+Cisplatin 80mg/m2 D1(or D1-3), 3-week chemotherapy for 3 cycles. After radiation, patients receive adjuvant chemotherapy Paclitaxel 135mg/m2 D1+Cisplatin 80mg/m2 D1(or D1-3), 3-week chemotherapy for 3 cycles.
  Arms: Standard-dose IMRT

SUMMARY:
Radiotherapy is an important treatment for initial distant metastases nasopharyngeal carcinoma. Total dose and fraction size are important prognostic factors for survival, although to our knowledge the optimal model has not been well determined to date. The purpose of this clinical trial is to investigate the optimal radiation dose to investigate the feasibility of decreasing the total dose and increasing the fraction size with the objective of achieving a better balance between local control and severe late complications. for initial distant metastases nasopharyngeal carcinoma with definitive radiotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if hypofractionated with a smaller total dose radiation is not inferior to standard-dose radiation in progression-free survival for initial distant metastases nasopharyngeal carcinoma .

SECONDARY OBJECTIVES:

I. To evaluate if hypofractionated with a low total dose radiation is not inferior to standard-dose radiation in overall survival and locoregional failure-free survival for initial distant metastases nasopharyngeal carcinoma II. To evaluate if hypofractionated with a low total dose radiation with chemotherapy decrease treatment-related toxicities

OUTLINE:

Patients are randomized to one of the two treatment arms

ARM 1: Patients receive hypofractionated with a low total dose radiation with induced chemotherapy and adjuvant chemotherapy.Hypofractionated dose IMRT: GTVnx 60Gy, GTVnd 60Gy, PTV1 50Gy and PTV2 45Gy in 25 fractions, 5 days/week.

Induced chemotherapy: Paclitaxel 135mg/m2 D1+Cisplatin 75mg/m2 D1(or D1-3), 3-week chemotherapy for 3 cycles. After radiation, patients receive adjuvant chemotherapy Paclitaxel 135mg/m2 D1+Cisplatin 75mg/m2 D1(or D1-3), 3-week chemotherapy for 3 cycles.

ARM 2: Patients receive standard-dose radiation with concurrent chemotherapy. Standard-dose IMRT: GTVnx 69.69Gy, GTVnd 60-68Gy, PTV1 59.4Gy and PTV2 54Gy in 33 fractions, 5 days/week.

Induced chemotherapy: Paclitaxel 135mg/m2 D1+Cisplatin 75mg/m2 D1(or D1-3), 3-week chemotherapy for 3 cycles. After radiation, patients receive adjuvant chemotherapy Paclitaxel 135mg/m2 D1+Cisplatin 75mg/m2 D1(or D1-3), 3-week chemotherapy for 3 cycles.

After completion of study therapy, patients are followed up every 3-4 months for 2 years, then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with newly histologically confirmed non-keratinizing (according to WHO histologically type) Tumor staged as any T or any N with M (according to the 8th AJCC edition).
2. No pregnant female
3. Age between 18-70
4. Normal complete blood count level (hemoglobin >10 g/dL, white blood cells ≥4000/μL, platelets ≥100 000/μL)
5. Normal hepatic functions (serum total bilirubin ≤1.6 mg/dL, serum transminase < 2.5 times higher than upper limit)
6. Normal renal function (serum creatinine ≤1.5 mg/dL, creatinine clearance ≥60 mL/min)
7. Karnofsky performance status (KPS) score of at least 70
8. Without radiotherapy or chemotherapy
9. Patients must give signed informed consent

Exclusion Criteria:

1. Other or mixed pathological type
2. age > 70 years or <18 years
3. Prior chemotherapy, radiation, surgical resection or target therapy of the primary tumor;
4. Significant medical or psychiatric illnesses that in the physician's judgment (uncontrolled coronary heart disease, cardiomyopathy and/or heart failure requiring hospitalization. Uncontrolled hypertension or history of myocardial infarction within one year. Uncontrolled diabetes mellitus. Acute bacterial or fungal infection requiring intravenous antibiotics;
5. Refused to sign informed consent form
6. Concurrent pregnancy or lactation
7. History of a second malignancy other than nasopharyngeal carcinoma

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-07-13 (Actual); Primary Completion 2020-06-10 (Actual); Study Completion 2022-04-10 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | 2 years
  The time from the first day of therapy to locoregional relapse, distant relapse or tumor-related death

SECONDARY OUTCOMES:
Overall survival | 2 years
  The time from the first day of therapy to death or last follow-up.
Locoregional relapse-free survival | 2 years
  The time from the first day of treatment to the time of first locoregional relapse
Distant metastasis-free survival | 2 years
  The time from the first day of treatment to the time of first distant metastasis

CONTACTS AND LOCATIONS:
Overall Officials: Wei Jiang, Ph.D., Study Director — Guilin Medical University, China
Locations (3):
- China (3):
  - Guangxi Naxishan Hospital, Guilin
  - Linshan people's hospital, Linshan
  - Wuzhou Red Cross Hospital, Wuzhou

REFERENCES:
- [Derived] Liu J, Zhang B, Su Y, Qin G, Kong X, Mo Y, Zhang R, Jiang W. Hypofractionated radiotherapy compared with conventionally fractionated radiotherapy to treat initial distant metastases in nasopharyngeal carcinoma: A multicenter, prospective, randomized, phase II trial. Radiother Oncol. 2023 Oct;187:109815. doi: 10.1016/j.radonc.2023.109815. Epub 2023 Jul 20. PMID 37480994